CLINICAL TRIAL: NCT05878639
Title: Evaluate Lactulose for Bowel Preparation in Patients With Inflammatory Bowel Disease
Brief Title: Efficacy and Safety of Lactulose for Bowel Preparation in Patients With Inflammatory Bowel Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SAHoWMU-CR2023-01-104
Record Dates: First submitted 2023-05-10; First posted 2023-05-26 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: IBD
Keywords: colonoscopy; polyethylene glycol; IBD; bowel preparation; lactulose
MeSH Terms: interventions — Polyethylene Glycols

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients take Lactulose for bowel preparation (Experimental): Patients take Lactulose for bowel preparation.
  Interventions: Drug: 3 bottles of Lactulose oral solution
- Patients take 3L-polyethylene glycol for bowel preparation (Active Comparator): Patients take 3L-polyethylene glycol for bowel preparation
  .
  Interventions: Drug: 3L-polyethylene glycol

INTERVENTIONS:
Drug: 3 bottles of Lactulose oral solution — Patients will take lactulose for bowel preparation.
  Arms: Patients take Lactulose for bowel preparation
Drug: 3L-polyethylene glycol — Patients will take 3L-polyethylene glycol for bowel preparation.
  Arms: Patients take 3L-polyethylene glycol for bowel preparation

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy, safety and tolerability of lactulose in bowel preparation in IBD patients. The main question it aims to answer is: Does lactulose have better efficacy, safety and tolerability than 3L-PEG? Participants will be divided into PEG group or Lactulose group at a 1:1 ratio by a random number method. Each patient will get a leaflet provided by hospital introducing bowel preparation methods and diet restriction before bowel preparation. They will have bowel preparation with different drugs according to group. The grade of bowel cleansing will be assessed through the Boston Bowel Preparation Scale (BBPS). The tolerability, satisfaction and safety of the two bowel preparation methods will be assessed through the patients self-administered questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* All patients with confirmed IBD or suspected IBD for at least 3 months, aged between 16-75 years and requiring a colonoscopy are invited to participate in our study. The diagnosis of IBD is based on recognized standards, including clinical symptoms, endoscopy, radiology, pathology and surgical history.

Exclusion Criteria:

* Patients are excluded if they (1) are clinical active UC and CD, (2) are known or suspected gastrointestinal obstruction, bowel perforation, toxic colitis or megacolon, recent or active gastrointestinal bleeding, (3) are congestive heart failure, severe renal failure, (4) are severe dehydration or electrolyte disturbances, (5) are pregnant, (6) are allergic to PEG or Lactulose, (7) are diabetics, (8) are lactose or galactose intolerance, (9) refuse to participate in this study.

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2023-03-28 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
effective preparation rate | 5 minutes before the colonoscopy ends
  Boston Bowel Preparation Scale (BBPS) >= 6 with a partial score >= 2 in each colon segment
incidence of adverse events | 2 hours after having bowel preparation
  incidence of adverse events in each group
taste score evaluated by patients | 2 hours after having bowel preparation
  Five-point scale is used to evaluate taste (very bad, bad, moderate, good, very good)

SECONDARY OUTCOMES:
effects of bowel preparation drugs on liver function | 2 hours after having bowel preparation
  total protein, albumin, bilirubin, alanine aminotransferase
effects of bowel preparation drugs on serum electrolyte | 2 hours after having bowel preparation
  sodium, potassium, chloride

CONTACTS AND LOCATIONS:
Overall Officials: Lin Daopo, Study Director — Department of Gastroenterology, The Second Affiliated Hospital of Wenzhou Medical University
Locations (1):
- The Second Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No